CLINICAL TRIAL: NCT05245825
Title: Effect of Flaxseed Supplementation on Glycemic Control in Prediabetic Adults
Brief Title: Flaxseed Supplementation in Prediabetic Adults (LINAPRED)
Acronym: LINAPRED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, Gabriela Macedo Ojeda, Professor researcher A, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI-01721
Record Dates: First submitted 2022-01-10; First posted 2022-02-18 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Prediabetic State
Keywords: Flax; Flaxseed; Linseed; Linum usitatissimum; Glycemic Control; Glycated Hemoglobin; Hemoglobin A1c; Glucose Tolerance Test; Blood glucose; Insulin resistance
MeSH Terms: conditions — Prediabetic State; Insulin Resistance | interventions — Linseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flaxseed and dietary plan (Experimental): 30 g of ground flaxseed daily and a dietary plan
  Interventions: Other: Flaxseed
- Control (Other): Dietary plan controlled in alpha-linolenic acid consumption
  Interventions: Other: Dietary plan

INTERVENTIONS:
Other: Flaxseed — A total of 30 g of ground flaxseed per day divided into two portions of 15 grams each, subjects will be asked to take 15 g in the morning and 15 g in the night dissolved in 400 ml of water. They will receive a dietary plan with a distribution of 20-30% of protein, 25-30% of lipids, and 40 to 45% of carbohydrates.
  Arms: Flaxseed and dietary plan
Other: Dietary plan — Dietary plan with a distribution of 20-30% of protein, 25-30% of lipids, and 40 to 45% of carbohydrates, controlled consumption of alpha-linolenic acid (no more than 6.8 g/day, the amount provided by 30 g of flaxseed).
  Arms: Control

SUMMARY:
Prediabetes is the term used to describe the condition where blood glucose level is higher than normal but lower than the diagnosis criteria of type 2 diabetes mellitus (T2DM). This condition confers a high risk for the development of T2DM and other diseases. Prediabetes could be reversible with lifestyle modifications, which include medical-nutrition therapy. Within these modifications, a healthy diet high in fiber and sources of alpha-linolenic acid is recommended. Flaxseed is a seed that is considered a functional food because it can provide health benefits due to its high content of fiber, alpha-linolenic acid, and lignans, these components could improve glycemic control in prediabetes patients by different mechanisms. The purpose of this study is to assess the effect of flaxseed on glycemic control in prediabetic adults.

DETAILED DESCRIPTION:
Prediabetes is a condition that increases the risk of T2DM and other diseases, its prevalence increases year after year despite being a reversible condition through lifestyle changes, diet, and medication. Therefore, it is important to find new strategies that, together with the known treatments, help to improve glycemic control in people with prediabetes and thus their risk of developing TDM2. Among these strategies may be the consumption of flaxseed, one of the main sources of alpha-linolenic acid (ALA), an omega-3 fatty acid, lignans, and fiber.

This open-label randomized clinical trial will include, prior informed consent, 96 men and women with prediabetes, subjects will be allocated in two groups, the intervention group or the control group. The intervention group will receive 30 g per day of ground flaxseed dissolved in water, (15 g in the morning and 15 g in the night), they will also be provided with a dietary plan. The Control group will not receive any supplementation, only a dietary plan controlled in alpha-linolenic acid.

The intervention will last 12 weeks; during this time, all patients will be scheduled every 2 weeks for follow-up visits. During the follow-up visits, subjects will be evaluated for changes in gastrointestinal symptoms, and adherence to supplementation, which will be assessed by a daily record, and the return of empty or unopened bags of flaxseed.

Every month, all subjects will undergo anthropometric, clinical, dietary, and biochemical evaluations that include measurements of body weight, body composition, waist, and hip circumferences, blood pressure, physical activity, quality of food intake, dietary intake, fasting plasma glucose, hemoglobin A1C, insulin, LDL-C, HDL-C, triglycerides, and total cholesterol; an oral glucose tolerance test will be performed at baseline and the end of the study to each subject.

At the end of the study, the obtained information will be shared with the scientific community to provide a possible food-based strategy for prediabetic adults in addition to the already known prediabetes treatment. All participants of the study will be beneficiated with free nutritional, anthropometric, and biochemical assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to participate in the study once they have read and signed the informed consent
* Men and women
* Fasting glucose levels between 100 and 125 mg/dl
* Age 30-59 years
* Stable weight in the last 3 months (no more than 5% weight change)

Exclusion Criteria:

* Fasting glucose <100 and >125 mg/dl
* Anemia
* Consumption of drugs that may modify glucose levels
* Consumption of flaxseed, chia, or omega-3, three months before the study
* Alternative diets (vegetarian, vegan, ketogenic, etc.)
* Pregnancy and breastfeeding
* Allergy or intolerance to flaxseed

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-11-20 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Fasting plasma glucose | 12 weeks
  Changes in plasma glucose concentration after the intervention (mg/dL)
2h-plasma glucose | 12 weeks
  Changes in 2h-plasma glucose concentration after an oral glucose tolerance test after the intervention (mg/dL)
Hemoglobin A1C | 12 weeks
  Changes in hemoglobin A1C after the intervention (%)

SECONDARY OUTCOMES:
Insulin | 12 weeks
  Changes in insulin concentration after the intervention (mUI/L)
Insulin resistance | 12 weeks
  Changes in insulin resistance after intervention assessed by the Homeostasis Model Assessment of Insulin Resistance (HOMA-IR), calculated using insulin and fasting plasma glucose concentrations
Lipid profile | 12 weeks
  Changes in total cholesterol, HDL-C, LDL-C, and triglycerides concentrations after the intervention (mg/dL)
Body Weight | 12 weeks
  Changes in body weight after the intervention (kg)
Body composition | 12 weeks
  Changes in body fat and muscle percentage after the intervention (%)
Waist and hip circumferences | 12 weeks
  Changes in waist and hip circumferences after the intervention (cm)
Blood pressure | 12 weeks
  Changes in systolic and diastolic blood pressure after the intervention (mmHg)
Physical activity level | 12 weeks
  Changes in total physical activity in METs-min/week assessed by the International Physical Activity Questionnaire - Short Form after the intervention
Food intake quality | 12 weeks
  Changes in food intake quality after the intervention assessed by the Mini-Survey to Evaluate Food Intake Quality (Mini-ECCA v.2)
Dietary ingestion | 12 weeks
  Changes in carbohydrate, protein, and fat ingestion after the intervention (g)
Stool classification | 12 weeks
  Changes in stool consistency will be assessed with The Bristol Stool Form Scale (BSFS) after the intervention.
  BSFS classifies stool into one of 7 stool types ranging from type 1 (hard lumps) to type 7 (watery), stool types 1 and 2 will be considered as constipation, stool types 5, 6, and 7 as diarrhea, and Stool types 3 and 4 as normal

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Macedo Ojeda, PhD, Study Director — University of Guadalajara
Locations (1):
- Universidad de Guadalajara (CUCS), Guadalajara, Jalisco, Mexico